CLINICAL TRIAL: NCT04911751
Title: A Phase 2, Double-Blind, Randomized, Placebo-Controlled, Study to Evaluate the Efficacy and Safety of KBL697 in Patients with Moderate Plaque Type Psoriasis
Brief Title: A Study to Investigate Efficacy and Safety of KBL697 in Patients with Moderate Plaque Type Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: KoBioLabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KBL-CURE-2020-02
Record Dates: First submitted 2021-05-09; First posted 2021-06-03 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Psoriatic Plaque
Keywords: microbiome; KBL697; Plaque psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low dose group (Experimental): 39 subjects for low dose group. 26 subjects on KBL697, 13 subjects on placebo.
  Interventions: Drug: KBL697
- High dose group (Experimental): 39 subjects for high dose group. 26 subjects on KBL697, 13 subjects on placebo.
  Interventions: Drug: KBL697

INTERVENTIONS:
Drug: KBL697 — 1 capsule BID of KBL697 or Placebo
  Arms: Low dose group
Drug: KBL697 — 5 capsules BID of KBL697 or Placebo
  Arms: High dose group

SUMMARY:
The study is designed to investigate efficacy and safety of KBL697 in patients with Moderate Plaque Type Psoriasis. KBL697 has been developed as a potential new treatment for Psoriatic Plaque.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 to 75 years (inclusive)
* Have a diagnosis of plaque type psoriasis for ≥ 6 months
* Must have chronic plaque type psoriasis of moderate severity
* All subjects must agree and commit to the use of a reliable contraceptive regimen.

Exclusion Criteria:

* Current diagnosis of forms of psoriasis other than chronic plaque type only
* Drug-induced psoriasis
* Other inflammatory skin disease that may confound the evaluation of plaque psoriasis
* Failed 2 or more systemic treatments for plaque psoriasis
* Medicinal shampoos that contain tar and/or salicylic acid within 2 weeks prior to Baseline Visit

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2024-10-07 (Actual)

PRIMARY OUTCOMES:
Psoriasis Area and Severity Index (PASI) | Baseline to Week 12
  Change from Baseline in PASI score

SECONDARY OUTCOMES:
Psoriasis Area and Severity Index (PASI) | Baseline to Weeks 2, 4 and 8
  Change from Baseline in PASI score
Psoriasis Area and Severity Index (PASI) -50 | Baseline to Week 12
  Percent of patients who achieved PASI-50
Psoriasis Area and Severity Index (PASI) -75 | Baseline to Week 12
  Percent of patients who achieved PASI-75
Physician's Global Assessment (PGA) | Baseline to Weeks 4, 8 and 12
  Change from Baseline in PGA score
Physician's Global Assessment (PGA) | Week 12
  Percent of patients who achieve PGA score of 0 or 1
Psoriasis-Affected Body Surface Area (BSA) | Baseline to Weeks 4, 8 and 12
  Change from Baseline in Psoriasis-Affected BSA
Safety measure through incidence of treatment-emergent adverse events (TEAEs) | Baseline to Week 16
  The number of patients experiencing TEAEs and number of individual TEAEs will be summarized among treatment arms, by system organ class (SOC) and PT. TEAEs will also be summarized among treatment arms, by severity and by relationship to study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Ira Thorla, Principal Investigator — Louisiana Dermatology Associates; Jose Cardona, Principal Investigator — Indago Research and Health Center; Jennifer Soung, Principal Investigator — Southern California Dermatology, Inc; James Krell, Principal Investigator — Total Skin and Beauty Dermatology Center; Paul Yamauchi, Principal Investigator — Clinical Science Institute; Ivette Espinosa-Fernandez, Principal Investigator — Revival Research Institute; Annika Smith, Principal Investigator — Westmead Hospital; Deirdre Murrell, Principal Investigator — Premier Specialist; Lynda Spelman, Principal Investigator — Veracity Clinical Trials Ltd; Samantha Eisman, Principal Investigator — Sinclair Dermatology
Locations (10):
- United States (6):
  - Total Skin and Beauty Dermatology Center, Birmingham, Alabama
  - Southern California Dermatology, Inc, Santa Ana, California
  - Clinical Science Institute, Santa Monica, California
  - Revival Research Institute, Doral, Florida
  - Indago Research and Health Center, Hialeah, Florida
  - Louisiana Dermatology Associates - Dermatology, Baton Rouge, Louisiana
- Australia (4):
  - Premier Specialist, Kogarah, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Veracity Clinical Trials Ltd, Woolloongabba, Queensland
  - Sinclair Dermatology, East Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No